CLINICAL TRIAL: NCT05722470
Title: Assessment of Prevalence of Eating Disorder Among Adolescents and it's Risk Factors
Brief Title: Eating Disorders Among Adolescents
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Rafek Mahmoud, Doctor, Assiut University
Other Study IDs: Eating disorders
Record Dates: First submitted 2023-01-16; First posted 2023-02-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: eating disorders — Assessment of eating disorders among adolescents

SUMMARY:
The aim of the present study is to evaluate the prevalence of eating disorder among adolescents. Also, to evaluate psychiatric comorbidity, sleep problems, alexithymia and emotion dysregulation associated with patients had eating disorders. In addition, to identify possible risk factors associated with eating disorder among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10 to 18 years old.
* Males and females are included.

Exclusion Criteria:

* - participants were previously diagnosed with any psychiatric disorder.

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Age between 10 and 18 years old Males and females
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
eating disorders among adolescents | baseline
  Assessment of prevalence of eating disorder among adolescents and it's risk factors